CLINICAL TRIAL: NCT06430476
Title: Ecological Momentary Intervention (EMI) as Augmentative Therapy for Depression in Clinical Sample in Hong Kong
Brief Title: EMI Therapy for Depression in Hong Kong
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EMI_depression
Record Dates: First submitted 2024-05-14; First posted 2024-05-28 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-04

CONDITIONS: Mild to Moderate Depression
Keywords: Depression; Ecological momentary intervention; Rumination; Hong Kong
MeSH Terms: conditions — Depression; Rumination Syndrome

STUDY DESIGN:
Intervention Model Description: EMA arm: participants will receive three ecological momentary assessment (EMA) prompts daily with the prompts spread out throughout the day. Within each prompt, participants will answer 14 questions regarding affect, suicidality, and rumination. Afterwards, they will be shown a video clip extracted from a popular and longstanding soap opera in Chinese that lasts between three to four minutes. Each prompt would take around 8 minutes to complete. In total, participants will complete 70 EMA prompts during the intervention period.
  EMI arm: participants will receive two EMA prompts and one EMI prompt daily. The EMA prompts would be identical to the ones in the EMA arm without the video clip at the end. The EMI prompt would contain an interactive task designed to counter ruminative thoughts.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: masking: Participants will be notified that they would engage in a diary recording activity for two weeks, but would be blinded to whether they were receiving the intervention or active control version. Participants will also be instructed not to reveal their exercise components (i.e., relaxation exercises or rumination exercises) to the trained research assistants, who will also be responsible for obtaining outcomes. Trained research assistents would assess outcomes and the principal investigator would randomise participants to the two conditions based on anonymised IDs. Treatment provided to participants as usual by their usual care providers (e.g., doctors) would not be notified about the randomisation conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMA (Active Comparator): Ecological momentary assessment (EMA) arm: participants will receive three ecological momentary assessment (EMA) prompts daily within three time blocks spread out throughout the day. Within each prompt, participants will answer 14 questions regarding affect, suicidality, and rumination. Afterwards, they will be shown a video clip extracted from a popular and longstanding soap opera in Chinese that lasts between three to four minutes. Each prompt would take around 8 minutes to complete. In total, participants will complete 70 EMA prompts during the intervention period.
  Interventions: Other: EMA
- EMI (Experimental): EMI arm: participants in this arm will receive two ecological momentary assessment (EMA) prompts and one econological momentary intervention (EMI) prompt daily. The EMA prompts would be identical to the ones in the EMA arm without the video clip at the end. The EMI prompt would contain an interactive task designed to counter ruminative thoughts. Examples of the interactive tasks include: mindfulness exercises (mindful walking), cognitive reappriasal, strengths recognition, etc. Each EMI prompt would last around 3-5 minutes.
  Interventions: Other: EMI

INTERVENTIONS:
Other: EMI — A phone-based intervention containing exercises meant to reduce ruminative thoughts carried out on an experience sampling platform m-Path
  Arms: EMI
Other: EMA — A phone-based exercise containing relaxation videos carried out on an experience sampling platform m-Path
  Arms: EMA

SUMMARY:
To determine if a two-week ecological momentary intervention (two EMA + one EMI daily) as augmentation to treatment as usual would reduce depressive symptoms, rumination levels, and functioning in subjects with mild to moderate depression, as compared to active controls receiving three EMA prompts daily.

DETAILED DESCRIPTION:
Background:

Major Depressive Disorder (MDD) is the leading contributors to disability-adjusted life years, with a burden comparable to that of cardiovascular disease. Among the core symptoms of MDD, rumination stands out as a particularly pernicious factor. Rumination is dysfunctional disturbing thinking; a maladaptive pattern of regulating thoughts and emotions characterized by a repetitive focus on negative thoughts, such as dwelling on negative memories and analyzing events without taking actions. Rumination amplifies negative cognitions and attenuates the effect of adapting problem-solving strategy, decreasing the motivation of patients to cope with stressful encounters and become more vulnerable to momentary low mood. Interventional strategies (such as Cognitive Bias Modification) targeting rumination involves increases one's ability to become aware of their own rumination and supporting them to adapt alternative thinking habits. Complementary techniques such as mindfulness and relaxation do not involve the reframing of negative thoughts but rather promote the acceptance of these thoughts, in this way, it allows one become more aware of distractions and repetitive past or future thinking events. The ESM, a structured self-report diary technique several times a day over a number of days using mobile devices zooming in on the micro-level of experience and behavior, presents a novel and promising approach to accurately track symptoms and experience by minimizing recall bias and capturing the natural fluctuations of symptom on a more immediate, granular level. The ESM-derived intervention (ESM-I), uses personalized mobile feedback to effectively treat depressive symptoms. Importantly, increasing evidence from randomised controlled trials (RCTs) have shown ESM-I as effective means to augment interventions in depression. While improving rumination is key the core depression symptom, ESM-I has yet to specifically target rumination, and the mechanisms by which ESM-I exert therapeutic effects warrant further investigation.

Objectives:

Our study aims to investigate the efficacy of a newly developed smartphone based 2-week Ecological Momentary Intervention (EMI) in comparison with an active control group receiving only ESM, as an innovative, online-based, accessible, and augmentative treatment for depression. This intervention is designed to be both timely and adaptive, targeting the core symptom of anhedonia in a clinical sample within Hong Kong.

Design:

This is a single-center, randomized, double-blind, sham-controlled trial with three assessment time points: Baseline (T0), post-intervention (T1) and 1-month post-intervention (T2).

Ecological Momentary Assessment (EMA): After providing informed consent, participants will install the "m-path" smartphone-based application, which is an open-source ESM program developed by KU Leuven. Following a briefing and practise run, participants will be randomly prompted within designated 3-hour blocks three times daily to complete a 5-minute questionnaire assessing their momentary affect, rumination levels, and suicidality, using visual analogue scales ranging from 0 (lowest) to 100 (highest). There will be 14 EMA questions covering affect (8 questions), suicidality (2 questions), and rumination (4 questions).

Ecological Momentary Intervention (EMI): Embedded within the last EMA survey, the EMI arm will include interactive tasks when a participant's computed rumination score (i.e., mean score of the four EMA rumination questions) reaches above the 80th percentile of their own cumulative score, or if the raw rumination score reach above 70 out of 100. The intervention comprises of short exercises (most can be completed within 1-3 minutes) rooted in cognitive bias modification (CBM) techniques. Participants will interact with instructions and multimedia formats based on CBM module framework based on reflection / brooding. Participants will continue treatment with their psychiatrists who will be blinded to group allocation.

Variables:

* Hamilton Depression Rating Scale (HDRS)
* Montgomery-Åsberg Depression Rating Scale (MADRS)
* Social and Occupational Functioning Assessment scale (SOFAS)
* Role Functioning Scale (RFS)
* Global Functioning: Social Scale and Role Scale
* Short Form Health Survey (SF-12)
* General Self Efficacy Scale
* Rumination Response Scale (RRS)
* System Usability Scale - Chinese version
* Beck Scale for Suicidal Ideation

ELIGIBILITY:
Inclusion Criteria:

* Aged 16-65 years
* Cantonese-speaking ethnic Chinese
* Diagnosis of major depressive episode (MDE) established by the Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorder 5th Edition (DSM-V)
* 17-item Hamilton Depression Rating Scale (HDRS) ≥ 14 at screening and at baseline (i.e. moderate to severe depression)
* Having a smartphone with Internet access and iOS or Android operating system.

Exclusion Criteria:

* Patients who could not read Chinese, are unable to provide informed consents
* Comorbid with other Axis I diagnoses (especially schizoaffective disorder)
* With an unstable medical condition or current substance abuse
* Have a score of ≥4 on any one of the three items on Positive and Negative Syndrome Scale (P1 Delusion, P2 Conceptual disorganization, P3 Hallucination)
* Marked risk of self-harm or suicide that could not be safely managed in an outpatient clinic setting
* Currently receiving any other weekly psychosocial therapy
* Unable to use a smartphone-based application due to cognitive impairment or learning disability or inadequate vision.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-06-30 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Ecological Momentary Assessment (EMA) outcomes | During intervention
  Average score among the following aspects: positive and negative affect (four questions each), active and passive suicidality (one question each), rumination (four questions); score ranges from 0 (minimal) to 100 (maximum), with a higher score indicating a greater value of measured aspect.
Montgomery-Åsberg Depression Rating Scale (MADRS) | T0 (baseline); T1 (immedately after intervention); T2 (one-month after intervention follow-up)
  Measuring change in depressive symptoms; score ranges from 0 (minimum) to 60 (maximum); higher score indicates more severe depressive symptoms.

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale (HDRS) - 17 items | T0 (baseline); T1 (immedately after intervention); T2 (one-month after intervention follow-up)
  Measuring depressive symptoms, score ranges from 0 (minimum) to 53 (maximum); higher score indicates more severe depressive symptoms.
Social and Occupational Functioning Assessment scale (SOFAS) | T0 (baseline); T1 (immedately after intervention); T2 (one-month after intervention follow-up)
  Measures social and occupational functioning across work functioning, independent functioning, immediate and extended social network functioning; score ranges from 0 (minimum) to 100 (maximum), higher score indicates higher social and occupational functioning ability.
Role Functioning Scale (RFS) | T0 (baseline); T1 (immedately after intervention); T2 (one-month after intervention follow-up)
  Measures role functioning in four areas: work productivity, independent living, immediate and extended social network relationships; score ranges from 0 (minimum) to 7 (maximum) on each aspect, higher score indicates better role functioning
Global Functioning: Social Scale and Role Scale | T0 (baseline); T1 (immedately after intervention); T2 (one-month after intervention follow-up)
  Measures social and role functioning; score ranges from 1 (minimum) to 10 (maximum); higher score indicates better social/role functioning
WHO-5 Well-being Index | T0 (baseline); T1 (immedately after intervention); T2 (one-month after intervention follow-up)
  Measures wellbeing at a primary care setting; score ranges from 0 (minimum) to 100 (maximum) and is calculated by summing the total score and multiply it by 4. Higher score indicates better wellbeing
General Self Efficacy Scale | T0 (baseline); T1 (immedately after intervention); T2 (one-month after intervention follow-up)
  Measures self-reported self-efficacy; score ranges from 10 (minimum) to 40 (maximum), with higher scores indicating more self-efficacy
Rumination Response Scale (RRS) | T0 (baseline); T1 (immedately after intervention); T2 (one-month after intervention follow-up)
  Measures self-reported rumination responses; score ranges from 10 (minimum) to 40 (maximum), with higher scores indicating higher levels of ruminative responses styles.
Beck Scale for Suicidal Ideation | T0 (baseline); T1 (immedately after intervention); T2 (one-month after intervention follow-up)
  Measures self-reported suicidal ideation; score ranges from 0 (minimum) to 38 (maximum), with higher scores indicating a greater risk of suicide.
System Usability Scale - Chinese version | T1 (immedately after intervention); T2 (one-month after intervention follow-up)
  to assess acceptability and feedback regarding conducting EMA and EMI on mPath platform; scores ranges from 10 (minimum) to 50 (maximum), with higher scores indicating higher perceived usability of the systems involved.
Clinical Global Impression Scale | T1 (immedately after intervention); T2 (one-month after intervention follow-up)
  Measures the severity of illness and global improvement following an intervention; scores ranges from 1 (normal/very much improved) to 7 (most severely ill/very much worse), with higher scores indicating worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Background] Morosini PL, Magliano L, Brambilla L, Ugolini S, Pioli R. Development, reliability and acceptability of a new version of the DSM-IV Social and Occupational Functioning Assessment Scale (SOFAS) to assess routine social functioning. Acta Psychiatr Scand. 2000 Apr;101(4):323-9. PMID 10782554
- [Background] Wang, Y., Lei, T., & Liu, X. (2020). Chinese System Usability Scale: Translation, Revision, Psychological Measurement. International Journal of Human-Computer Interaction, 36(10), 953-963. https://doi.org/10.1080/10447318.2019.1700644
- [Background] American Psychiatric Association. (2013). Diagnostic and statistical manual of mental disorders (5th ed.). https://doi.org/10.1176/appi.books.9780890425596
- [Background] Mestdagh M, Verdonck S, Piot M, Niemeijer K, Kilani G, Tuerlinckx F, Kuppens P, Dejonckheere E. m-Path: an easy-to-use and highly tailorable platform for ecological momentary assessment and intervention in behavioral research and clinical practice. Front Digit Health. 2023 Oct 18;5:1182175. doi: 10.3389/fdgth.2023.1182175. eCollection 2023. PMID 37920867
- [Background] Devilly GJ, Borkovec TD. Psychometric properties of the credibility/expectancy questionnaire. J Behav Ther Exp Psychiatry. 2000 Jun;31(2):73-86. doi: 10.1016/s0005-7916(00)00012-4. PMID 11132119